CLINICAL TRIAL: NCT05720949
Title: Genicular Nerve Blocks for Arthroscopic Anterior Cruciate Knee Surgery: a Randomized Controlled Trial
Brief Title: Genicular Nerve Blocks for Anterior Cruciate Ligament Knee Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022-1962
Record Dates: First submitted 2023-01-18; First posted 2023-02-09 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2024-12

CONDITIONS: ACL; Anterior Cruciate Ligament Injuries
Keywords: ACL; Genicular nerve block; Anterior Cruciate Ligament Injuries; Opioid Consumption
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Bupivacaine; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Double blind randomized control trail
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient, research assistants, and biostatisticians are blinded to whether the patient was randomized to the control or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 - Control (No Intervention): Patients randomized to this group will receive an adductor canal block (ACB) and Infiltration between the Popliteal Artery and Capsule of the Knee (IPACK) nerve block.
- Group 2 - Intervention (Experimental): Patients randomized to this group will receive an adductor canal block (ACB), Infiltration between the Popliteal Artery and Capsule of the Knee (IPACK) nerve block, and the genicular nerve block (intervention).
  The genicular nerve block is a total of 20cc of 0.25% bupivacaine with 2mg of preservative free dexamethasone applied to the superomedial genicular nerve, superolateral genicular nerve, inferomedial genicular nerve, and nerve to vastus intermedius.
  Interventions: Drug: Genicular Nerve Block with bupivacaine and preservative free dexamethasone

INTERVENTIONS:
Drug: Genicular Nerve Block with bupivacaine and preservative free dexamethasone — A genicular nerve block is a peripheral nerve block that temporarily anesthetizes the sensory terminal branches innervating the knee joint by injecting local anesthesia. This results in anesthesia of the anterior compartment of the knee.
  The genicular nerve block consists of 20cc of 0.25% bupivacaine with 2mg of preservative free dexamethasone and will be applied to the superomedial genicular nerve, superolateral genicular nerve, inferomedial genicular nerve, and nerve to vastus intermedius.
  Bupivacaine - Drug class: Sodium channel blocker
  Dexamethasone - Drug class: Glucocorticoid
  Other Names: Exparel; Ozurdex
  Arms: Group 2 - Intervention

SUMMARY:
The purpose of this randomized controlled trial is to assess a new analgesia regimen that includes the addition of genicular never blocks to our current standard regimen of peripheral nerve blocks, which includes an adductor canal block (ACB) and interspace between the popliteal artery and capsule of the posterior knee block (IPACK). The main questions it aims to answer are:

1. Does addition of genicular nerve blocks to standard peripheral block regimen significantly reduce the mean opioid consumption by 33% in the first 24 hours?
2. Does genicular nerve blocks reduce NRS pain scores?
3. Does genicular nerve blocks facilitate earlier discharge?
4. Does genicular nerve blocks last longer than 24 hours?
5. Does genicular nerve blocks improve pain management?

Eligible patients are those undergoing an anterior cruciate ligament repair at the Hospital for Special Surgery and participants will be randomized to receive the intervention (genicular nerve block) or the standard of care.

DETAILED DESCRIPTION:
Genicular nerve blocks have been shown to provide effective analgesia for chronic osteoarthritis knee pain. There are several publications supporting its use for chronic knee pain but there is a scarcity of literature in its use in the perioperative period. Recently, it has been shown to provide effective analgesia for total knee arthroplasty. This will be a novel application for it to be used for anterior cruciate ligament surgery. There are only a couple of prospective and retrospective studies that showed promising analgesic benefits for anterior cruciate ligament repairs. There are currently no randomized controlled trials published investigating the use of genicular nerve blocks for anterior cruciate ligament surgery.

Researching novel innovative motor-sparing and opioid-sparing peripheral nerve blocks for have been the focus of research. Studies have investigated the motor sparing benefits of the adductor canal block, the effective analgesic benefits of the IPACK block, the phrenic sparing benefits of the superior trunk block, and the analgesic benefits of the pericapsular nerve group block and lateral femoral cutaneous nerve. Genicular nerve blocks would be a potential additive block that may further enhance the recovery of patients undergoing knee surgeries, including unicondylar, total knee and anterior cruciate ligament repair patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80
* English speaking
* American Society of Anesthesiologists (ASA) I - III
* BMI < 35
* Scheduled for ambulatory arthroscopic unilateral anterior cruciate ligament repair surgery with bone tendon bone autograft

Exclusion Criteria:

* History of chronic pain syndromes
* Chronic opioid use (daily morphine milligram equivalents > 30 mg for at least 3 months)
* Contraindication to peripheral nerve blocks
* Contraindication to neuraxial anesthesia
* History of peripheral neuropathy or pre-existing neurological deficits
* Psychiatric or cognitive disorder that prohibit patient from following study protocol
* Allergy to local anesthetic or study medications
* Multi-ligament surgery
* History of substance abuse
* Infection at the site of injection
* diagnoses of Type I or Type II diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jashvant Poeran, MD/PhD, Study Director — Hospital for Special Surgery, Department of Anesthesiology; David H Kim, MD, Principal Investigator — Hospital for Special Surgery, Department of Anesthesiology
Locations (1):
- HSS Sports Medicine Institute West Side, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data with other researchers.

REFERENCES:
- [Background] Conger A, Gililland J, Anderson L, Pelt CE, Peters C, McCormick ZL. Genicular Nerve Radiofrequency Ablation for the Treatment of Painful Knee Osteoarthritis: Current Evidence and Future Directions. Pain Med. 2021 Jul 25;22(Suppl 1):S20-S23. doi: 10.1093/pm/pnab129. PMID 34308957
- [Background] Rambhia M, Chen A, Kumar AH, Bullock WM, Bolognesi M, Gadsden J. Ultrasound-guided genicular nerve blocks following total knee arthroplasty: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2021 Oct;46(10):862-866. doi: 10.1136/rapm-2021-102667. Epub 2021 Jul 14. PMID 34261807
- [Background] Caldwell GL Jr, Selepec MA. Reduced Opioid Use After Surgeon-Administered Genicular Nerve Block for Anterior Cruciate Ligament Reconstruction in Adults and Adolescents. HSS J. 2019 Feb;15(1):42-50. doi: 10.1007/s11420-018-09665-9. Epub 2019 Jan 28. PMID 30863232
- [Background] Gruskay JA, Pearce SS, Ruttum D, Conrad ES 3rd, Hackett TR. Surgeon-Administered Anterolateral Geniculate Nerve Block as an Adjunct to Regional Anesthetic for Pain Management Following Anterior Cruciate Ligament Reconstruction. Arthrosc Tech. 2022 Jan 20;11(1):e1-e6. doi: 10.1016/j.eats.2021.08.034. eCollection 2022 Jan. PMID 35127422
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Background] Kim DH, Beathe JC, Lin Y, YaDeau JT, Maalouf DB, Goytizolo E, Garnett C, Ranawat AS, Su EP, Mayman DJ, Memtsoudis SG. Addition of Infiltration Between the Popliteal Artery and the Capsule of the Posterior Knee and Adductor Canal Block to Periarticular Injection Enhances Postoperative Pain Control in Total Knee Arthroplasty: A Randomized Controlled Trial. Anesth Analg. 2019 Aug;129(2):526-535. doi: 10.1213/ANE.0000000000003794. PMID 30234517
- [Background] Kim DH, Lin Y, Beathe JC, Liu J, Oxendine JA, Haskins SC, Ho MC, Wetmore DS, Allen AA, Wilson L, Garnett C, Memtsoudis SG. Superior Trunk Block: A Phrenic-sparing Alternative to the Interscalene Block: A Randomized Controlled Trial. Anesthesiology. 2019 Sep;131(3):521-533. doi: 10.1097/ALN.0000000000002841. PMID 31283740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between January 12, 2023 and November 25, 2024 in the preoperative holding area of the Hospital for Special Surgery West Side Ambulatory Surgery Center.
Groups:
- Group 2 - Intervention: Patients randomized to this group will receive an adductor canal block (ACB), Infiltration between the Popliteal Artery and Capsule of the Knee (IPACK) nerve block, and the genicular nerve block (intervention).
  The genicular nerve block is a total of 20cc of 0.25% bupivacaine with 2mg of preservative free dexamethasone applied to the superomedial genicular nerve, superolateral genicular nerve, inferomedial genicular nerve, and nerve to vastus intermedius.
  Genicular Nerve Block with bupivacaine and preservative free dexamethasone: A genicular nerve block is a peripheral nerve block that temporarily anesthetizes the sensory terminal branches innervating the knee joint by injecting local anesthesia. This results in anesthesia of the anterior compartment of the knee.
  The genicular nerve block consists of 20cc of 0.25% bupivacaine with 2mg of preservative free dexamethasone and will be applied to the superomedial genicular nerve, superolateral genicular nerve, inferomedial genicular nerve, and nerve to vastus intermedius.
  Bupivacaine - Drug class: Sodium channel blocker
  Dexamethasone - Drug class: Glucocorticoid
Period: Overall Study
Arm/Group | Group 1 - Control | Group 2 - Intervention
Started | 96 | 96
Completed | 85 | 82
Not Completed | 11 | 14
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 11 | 13

BASELINE CHARACTERISTICS:
Population: Total number of participants who were enrolled and randomized for whom baseline characteristics were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Control | Group 2 - Intervention | Total
Number analyzed (Participants) | 96 | 95 | 191
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: One patient withdrew in the intervention group.
  years | 26.51 [21.90 to 30.08] | 26.03 [22.21 to 29.72] | 26.48 [22.10 to 29.84]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient withdrew in the intervention group.
  Participants
    Female | 39 | 37 | 76
    Male | 57 | 58 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One patient withdrew in the intervention group.
  Participants
    Hispanic or Latino | 12 | 13 | 25
    Not Hispanic or Latino | 81 | 80 | 161
    Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One patient withdrew from the intervention group.
  Participants
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 17 | 14 | 31
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 5 | 2 | 7
    White | 59 | 63 | 122
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 13 | 16 | 29
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] — Population: One patient withdrew from the intervention group.
  kg/m^2 | 23.95 [22.12 to 25.87] | 24.58 [22.88 to 28.01] | 24.27 [22.31 to 26.78]

OUTCOME MEASURES:

1. Primary Outcome: Mean Opioid Consumption at 24 Hours
Description: Intravenous and Oral opioid consumption at 24 hours after recovery room entry will be recorded.
  The average consumption will be reported in morphine milligram equivalents.
Time Frame: Post-operative care unit (PACU) arrival time to 24 hours
Population: Participants were lost to follow up in both groups.
Measure: Mean (Full Range); unit: morphine milligram equivalents
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 89 | 86
morphine milligram equivalents | 21.5 [0 to 67.5] | 19.9 [0 to 97.5]
Statistical Analysis 1: Comparison: Group 1 - Control vs Group 2 - Intervention; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Opioid Consumption
Description: Opioid consumption up to 168 hours after surgery will be recorded from the medical record and patient reported phone calls
  Opioid consumption in morphine milligram equivalents will be calculated and reported for each time point.
Time Frame: PACU(PACU arrival time to removal from board), 48,72,96,168 hours after time zero (PACU arrival time)
Population: At each time point, patients were lost to follow up.
Measure: Median (Full Range); unit: morphine milligram equivalents
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 96 | 95
morphine milligram equivalents
  PACU | 7.5 [0 to 30] | 7.5 [0 to 30]
  48 hours: number analyzed (Participants) | 88 | 83
  48 hours | 15 [0 to 45.0] | 11.25 [0 to 60.0]
  72 hours: number analyzed (Participants) | 87 | 83
  72 hours | 7.5 [0 to 52.5] | 0 [0 to 60.0]
  96 hours: number analyzed (Participants) | 86 | 82
  96 hours | 0 [0 to 33.75] | 0 [0 to 60.0]
  168 hours: number analyzed (Participants) | 85 | 82
  168 hours | 0 [0 to 15.0] | 0 [0 to 22.5]
Statistical Analysis 1: Comparison: Group 1 - Control vs Group 2 - Intervention; PACU; Test type: Superiority; p = 0.037, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group 1 - Control vs Group 2 - Intervention; 72 hours; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group 1 - Control vs Group 2 - Intervention; 96 hours; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Group 1 - Control vs Group 2 - Intervention; 168 hours; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Numeric Rating Scale (NRS) Pain Scores
Description: Patient scores at rest and with movement will be recorded. Scale of 0 to 10, with 0 meaning "no pain" and 10 meaning "worst pain imaginable". Lower score means less pain, higher score means greater pain.
Time Frame: PACU (60 minutes after PACU arrival time), 24,48,72,96,168 hours after time zero (PACU arrival time)
Population: At each time point, patients were lost to follow up.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 96 | 95
score on a scale
  PACU-rest | 3 [0 to 8] | 2 [0 to 8]
  PACU-movement | 4 [0 to 8] | 2.5 [0 to 8]
  24 hours-rest: number analyzed (Participants) | 89 | 86
  24 hours-rest | 3 [0 to 10] | 3 [0 to 9]
  24 hours-movement: number analyzed (Participants) | 89 | 86
  24 hours-movement | 5 [0 to 10] | 5 [0 to 10]
  48 hours-rest: number analyzed (Participants) | 88 | 83
  48 hours-rest | 3 [0 to 10] | 3 [1 to 8]
  48 hours-movement: number analyzed (Participants) | 88 | 83
  48 hours-movement | 5 [0 to 10] | 5 [0 to 10]
  72 hours-rest: number analyzed (Participants) | 86 | 82
  72 hours-rest | 3 [0 to 9] | 2 [0 to 7]
  72 hours-movement: number analyzed (Participants) | 86 | 82
  72 hours-movement | 4 [0 to 9] | 4 [0 to 9]
  96 hours-rest: number analyzed (Participants) | 86 | 82
  96 hours-rest | 2 [0 to 9] | 2 [0 to 7]
  96 hours-movement: number analyzed (Participants) | 86 | 82
  96 hours-movement | 4 [0 to 10] | 4 [1 to 8]
  168 hours-rest: number analyzed (Participants) | 85 | 82
  168 hours-rest | 1 [0 to 9] | 1 [0 to 7]
  168 hours-movement: number analyzed (Participants) | 85 | 82
  168 hours-movement | 3 [0 to 9] | 3 [0 to 8]
Statistical Analysis 1: Comparison: Group 1 - Control vs Group 2 - Intervention; PACU-rest; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 - Control vs Group 2 - Intervention; PACU-movement; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 hours-rest; Test type: Superiority; p = 0.2, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 hours-movement; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours-rest; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours-movement; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Group 1 - Control vs Group 2 - Intervention; 72 hours-rest; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Group 1 - Control vs Group 2 - Intervention; 72 hours-movement; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Group 1 - Control vs Group 2 - Intervention; 96 hours-rest; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Group 1 - Control vs Group 2 - Intervention; 96 hours-movement; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Group 1 - Control vs Group 2 - Intervention; 168 hours-rest; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Group 1 - Control vs Group 2 - Intervention; 168 hours-movement; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Cumulative Opioid Consumption
Description: Total opioid consumption will be recorded up to 96 hours after surgery.
Time Frame: sum of opioid used from 0-24 hours, 0-48 hours, and 0-72 hours, 0-96 hours post-operatively
Population: At each time point, patients were lost to follow up.
Measure: Median (Full Range); unit: morphine milligram equivalents
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 96 | 95
morphine milligram equivalents
  0-24 hours: number analyzed (Participants) | 89 | 86
  0-24 hours | 22.5 [0 to 67.5] | 15 [0 to 97.5]
  0-48 hours: number analyzed (Participants) | 88 | 83
  0-48 hours | 33.75 [0 to 105] | 30 [0 to 142.5]
  0-72 hours: number analyzed (Participants) | 87 | 83
  0-72 hours | 37.5 [0 to 142.5] | 37.5 [0 to 165]
  0-96 hours: number analyzed (Participants) | 86 | 82
  0-96 hours | 41.3 [0 to 168.75] | 45 [0 to 225]
Statistical Analysis 1: Comparison: Group 1 - Control vs Group 2 - Intervention; 0-24 hours; Test type: Superiority; p = 0.17, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 - Control vs Group 2 - Intervention; 0-48 hours; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group 1 - Control vs Group 2 - Intervention; 0-72 hours; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group 1 - Control vs Group 2 - Intervention; 0-96 hours; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Brief Pain Inventory
Description: This questionnaire will assess severity of pain, impact of pain on daily function, location of pain, medication intake, and amount of pain relief preoperatively and at 24 hours, 48 hours, 72 hours, 96 hours, and 168 hours after surgery.
  Questions are rated on a scale of 0 to 10, with 0 meaning "no pain/interference" and 10 meaning "pain as bad as you can imagine/completely interferes".
Time Frame: Pre-operatively, 24 hours, 48 hours, 72 hours, 96 hours, 168 hours post-operative
Population: At each time point, patients were lost to follow up.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 96 | 95
score on a scale
  Preoperative Worst Pain | 2 [0 to 10] | 2 [0 to 9]
  Preoperative Least Pain | 0 [0 to 7] | 0 [0 to 6]
  Preoperative Average Pain | 1 [0 to 8] | 1 [0 to 6]
  Preoperative Current Pain | 0 [0 to 8] | 0 [0 to 5]
  Preoperative Interference: number analyzed (Participants) | 91 | 91
  Preoperative Interference | 1.14 [0 to 6.86] | 1.14 [0 to 8.43]
  24 hours worst pain: number analyzed (Participants) | 89 | 86
  24 hours worst pain | 7 [2 to 10] | 7 [0 to 10]
  24 hours least pain: number analyzed (Participants) | 89 | 86
  24 hours least pain | 2 [0 to 9] | 2 [0 to 7]
  24 hours average pain: number analyzed (Participants) | 89 | 86
  24 hours average pain | 4 [0 to 10] | 3 [0 to 9]
  24 hours current pain: number analyzed (Participants) | 89 | 86
  24 hours current pain | 3 [0 to 10] | 3 [0 to 9]
  24 hours interference: number analyzed (Participants) | 84 | 81
  24 hours interference | 3.57 [0 to 8.57] | 3.07 [0 to 8]
  48 hours worst pain: number analyzed (Participants) | 88 | 83
  48 hours worst pain | 7 [0 to 10] | 6 [2 to 10]
  48 hours least pain: number analyzed (Participants) | 88 | 83
  48 hours least pain | 2 [0 to 10] | 2 [0 to 6]
  48 hours average pain: number analyzed (Participants) | 88 | 83
  48 hours average pain | 4 [0 to 10] | 4 [0 to 8]
  48 hours current pain: number analyzed (Participants) | 88 | 83
  48 hours current pain | 3 [0 to 10] | 3 [0 to 8]
  48 hours interference: number analyzed (Participants) | 83 | 79
  48 hours interference | 4.14 [0 to 8.71] | 3.86 [0 to 8.43]
  72 hours worst pain: number analyzed (Participants) | 87 | 83
  72 hours worst pain | 6 [0 to 10] | 6 [1 to 10]
  72 hours least pain: number analyzed (Participants) | 87 | 83
  72 hours least pain | 2 [0 to 8] | 1 [0 to 6]
  72 hours average pain: number analyzed (Participants) | 87 | 83
  72 hours average pain | 3 [0 to 8] | 3 [0 to 7]
  72 hours current pain: number analyzed (Participants) | 87 | 83
  72 hours current pain | 3 [0 to 9] | 2 [0 to 7]
  72 hours interference: number analyzed (Participants) | 83 | 81
  72 hours interference | 6 [0 to 10] | 5 [0 to 10]
  96 hours worst pain: number analyzed (Participants) | 86 | 82
  96 hours worst pain | 5 [0 to 10] | 5 [1 to 9]
  96 hours least pain: number analyzed (Participants) | 86 | 82
  96 hours least pain | 1 [0 to 8] | 1 [0 to 6]
  96 hours average pain: number analyzed (Participants) | 86 | 82
  96 hours average pain | 2 [0 to 9] | 3 [0 to 8]
  96 hours current pain: number analyzed (Participants) | 86 | 82
  96 hours current pain | 2 [0 to 9] | 2 [0 to 7]
  96 hours interference: number analyzed (Participants) | 84 | 81
  96 hours interference | 3.14 [0 to 8] | 2.86 [0 to 8.57]
  168 hours worst pain: number analyzed (Participants) | 85 | 82
  168 hours worst pain | 4 [1 to 10] | 4 [1 to 9]
  168 hours least pain: number analyzed (Participants) | 85 | 82
  168 hours least pain | 0 [0 to 8] | 0 [0 to 6]
  168 hours average pain: number analyzed (Participants) | 85 | 82
  168 hours average pain | 2 [0 to 9] | 2 [0 to 8]
  168 hours current pain: number analyzed (Participants) | 85 | 82
  168 hours current pain | 1 [0 to 9] | 1 [0 to 7]
  168 hours interference: number analyzed (Participants) | 82 | 81
  168 hours interference | 2.14 [0 to 6.14] | 2 [0 to 8.29]
Statistical Analysis 1: Comparison: Group 1 - Control vs Group 2 - Intervention; Preoperative Worst Pain; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 - Control vs Group 2 - Intervention; Preoperative Least Pain; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group 1 - Control vs Group 2 - Intervention; Preoperative Average Pain; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group 1 - Control vs Group 2 - Intervention; Preoperative Current Pain; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Group 1 - Control vs Group 2 - Intervention; Preoperative Interference; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 hours worst pain; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 hours least pain; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 hours average pain; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 hours current pain; Test type: Superiority; p = 0.21, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 hours interference; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours worst pain; Test type: Superiority; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours least pain; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours average pain; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours current pain; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours interference; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Group 1 - Control vs Group 2 - Intervention; 72 hours worst pain; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Group 1 - Control vs Group 2 - Intervention; 72 hours least pain; Test type: Superiority; p = 0.35, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Group 1 - Control vs Group 2 - Intervention; 72 hours average pain; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Group 1 - Control vs Group 2 - Intervention; 72 hours current pain; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Group 1 - Control vs Group 2 - Intervention; 72 hours interference; Test type: Superiority; p = 0.11, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Group 1 - Control vs Group 2 - Intervention; 96 hours worst pain; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Group 1 - Control vs Group 2 - Intervention; 96 hours least pain; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Group 1 - Control vs Group 2 - Intervention; 96 hours average pain; Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Group 1 - Control vs Group 2 - Intervention; 96 hours current pain; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Group 1 - Control vs Group 2 - Intervention; 96 hours interference; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Group 1 - Control vs Group 2 - Intervention; 168 hours worst pain; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Group 1 - Control vs Group 2 - Intervention; 168 hours least pain; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Group 1 - Control vs Group 2 - Intervention; 168 hours average pain; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney)
Statistical Analysis 29: Comparison: Group 1 - Control vs Group 2 - Intervention; 168 hours current pain; Test type: Superiority; p = 0.93, Wilcoxon (Mann-Whitney)
Statistical Analysis 30: Comparison: Group 1 - Control vs Group 2 - Intervention; 168 hours interference; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Patient Satisfaction With Pain Treatment
Description: Patient satisfaction will be assessed in the post-operative care unit (PACU), 24 hours, and 48 hours after surgery.
  Patients reported satisfaction for 3 subcategories: 1) Satisfaction with Pain Management, 2) Satisfaction with Being Informed and Involved with Decision Making, 3) Satisfaction with Care from Healthcare Team. Each subcategory had a scale of 0-10, with 0 being strongly dissatisfied and 10 being strongly satisfied.
Time Frame: From the time patient arrived in the post-operative care unit (PACU), at 24 hours, and at 48 hours post-operative
Population: At each time point, patients were lost to follow up.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 96 | 95
score on a scale
  PACU Satisfaction with Pain Management | 10 [0 to 10] | 10 [5 to 10]
  PACU Satisfaction with Being Informed and Involved with Decision Making | 10 [6 to 10] | 10 [4 to 10]
  PACU Satisfaction with Care from Healthcare Team | 10 [7 to 10] | 10 [8 to 10]
  24 Hours Satisfaction with Pain Management: number analyzed (Participants) | 89 | 86
  24 Hours Satisfaction with Pain Management | 9 [0 to 10] | 9.5 [5 to 10]
  24 hours Satisfaction with Being Informed and Involved with Decision Making: number analyzed (Participants) | 89 | 86
  24 hours Satisfaction with Being Informed and Involved with Decision Making | 10 [6 to 10] | 10 [4 to 10]
  24 hours Satisfaction with Care from Healthcare Team: number analyzed (Participants) | 89 | 86
  24 hours Satisfaction with Care from Healthcare Team | 10 [5 to 10] | 10 [6 to 10]
  48 Hours Satisfaction with Pain Management: number analyzed (Participants) | 88 | 83
  48 Hours Satisfaction with Pain Management | 9 [0 to 10] | 10 [5 to 10]
  48 hours Satisfaction with Being Informed and Involved with Decision Making: number analyzed (Participants) | 88 | 83
  48 hours Satisfaction with Being Informed and Involved with Decision Making | 10 [6 to 10] | 10 [4 to 10]
  48 hours Satisfaction with Care from Healthcare Team: number analyzed (Participants) | 88 | 83
  48 hours Satisfaction with Care from Healthcare Team | 10 [6 to 10] | 10 [6 to 10]
Statistical Analysis 1: Comparison: Group 1 - Control vs Group 2 - Intervention; PACU Satisfaction with Pain Management; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 - Control vs Group 2 - Intervention; PACU Satisfaction with Being Informed and Involved with Decision Making; Test type: Superiority; p = 0.028, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group 1 - Control vs Group 2 - Intervention; PACU Satisfaction with Care from Healthcare Team; Test type: Superiority; p = 0.032, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 Hours Satisfaction with Pain Management; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 hours Satisfaction with Being Informed and Involved with Decision Making; Test type: Superiority; p = 0.36, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 hours Satisfaction with Care from Healthcare Team; Test type: Superiority; p = 0.91, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 Hours Satisfaction with Pain Management; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours Satisfaction with Being Informed and Involved with Decision Making; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours Satisfaction with Care from Healthcare Team; Test type: Superiority; p = 0.59, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Duration of Analgesic Block
Description: To assess when the patient believe the analgesic block wore off and they regain sensation in their leg.
Time Frame: 24 hours and 48 hours post-operative
Population: At each time point, some patients were lost to follow up and some patients did not have feeling return yet.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 96 | 95
hours
  24 hours: number analyzed (Participants) | 53 | 42
  24 hours | 15.8 [5.03 to 22.65] | 13.825 [8.22 to 21.97]
  48 hours: number analyzed (Participants) | 78 | 70
  48 hours | 22.19 [10.92 to 35.77] | 25.05 [11.83 to 38.15]
Statistical Analysis 1: Comparison: Group 1 - Control vs Group 2 - Intervention; 24 hours; Test type: Superiority; p = 0.93, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 - Control vs Group 2 - Intervention; 48 hours; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Success of Adductor Canal Block
Description: Numbness in the saphenous distribution will be assessed in the PACU by an anesthesiologist or research assistant. This was measured on scale of 0-2, with 0 being no sensation, 1 being partial sensation, and 2 being full sensation.
Time Frame: Post-operative care unit (PACU)
Population: One patient was withdrawn from the intervention group. For one patient in the control group, data was not able to be obtained for success of adductor canal block.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 95 | 95
Participants
  Medial Calf: No sensation | 28 | 55
  Medial Calf: Partial sensation | 45 | 32
  Medial Calf: Full sensation | 22 | 8
  Lateral Calf: No sensation | 9 | 16
  Lateral Calf: Partial sensation | 41 | 61
  Lateral Calf: Full sensation | 45 | 18
  Dorsal Calf: No sensation | 11 | 7
  Dorsal Calf: Partial sensation | 27 | 58
  Dorsal Calf: Full sensation | 57 | 30
  Plantar Aspect: No sensation | 1 | 3
  Plantar Aspect: Partial sensation | 37 | 53
  Plantar Aspect: Full sensation | 57 | 39
Statistical Analysis 1: Comparison: Group 1 - Control vs Group 2 - Intervention; Medial Calf; Test type: Superiority; p = 0.0002, Chi-squared
Statistical Analysis 2: Comparison: Group 1 - Control vs Group 2 - Intervention; Lateral Calf; Test type: Superiority; p = 0.0002, Chi-squared
Statistical Analysis 3: Comparison: Group 1 - Control vs Group 2 - Intervention; Dorsal Calf; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 4: Comparison: Group 1 - Control vs Group 2 - Intervention; Plantar Aspect; Test type: Superiority; p = 0.027, Chi-squared

9. Secondary Outcome: Readiness for PACU Discharge
Description: The duration from PACU arrival time to recovery complete time.
  The time that it took for the patient to be discharged will be calculated and reported.
Time Frame: From the time the patient arrived in the post-operative care unit (PACU) arrival time to the time the patient is discharged(discharge ready time = recovery complete time) assessed up to 24 hours after surgery.
Population: One patient was withdrawn from the intervention group.
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 96 | 95
hours | 1.69 [0.1 to 3.3] | 1.67 [0.75 to 2.93]
Statistical Analysis 1: Comparison: Group 1 - Control vs Group 2 - Intervention; Test type: Superiority; p = 0.928, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Length of PACU Stay
Description: The duration from PACU arrival time to patient removed from board time.
  The time (in minutes) will be calculated and reported.
Time Frame: From the time the patient arrived in the post-operative care unit (PACU) arrival time to the time they leave the PACU assessed up to 24 hours after surgery.
Population: One patient was withdrawn from the intervention group.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 96 | 95
minutes | 125.5 [111.5 to 147.0] | 124.0 [109.0 to 146.0]
Statistical Analysis 1: Comparison: Group 1 - Control vs Group 2 - Intervention; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Adverse Events
Description: Incidence of neuropraxia (neurological symptoms over 3 days), local anesthetic systemic toxicity (LAST), and infection.
  The number of adverse events will be reported.
Time Frame: Post-operative care unit (PACU) arrival time up to 72 hours after the surgery
Population: One patient was withdrawn from the intervention group.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Control | Group 2 - Intervention
Number analyzed (Participants) | 96 | 95
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Follow ups occurred up to 7 days postoperatively.
Arm/Group | Group 1 - Control | Group 2 - Intervention
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/96
Other Adverse Events (participants affected / at risk) | 0/96 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT05720949/Prot_SAP_000.pdf